CLINICAL TRIAL: NCT06454045
Title: Evaluation of Platelet Aggregability in Patients With Previous Acute Myocardial Infarction or Concomitant Lower Extremity Peripheral Artery Disease
Status: Active, not recruiting | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Jose Carlos Nicolau, Professor, University of Sao Paulo
Other Study IDs: SDC: 5794/24/005
Record Dates: First submitted 2024-05-15; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease; Peripheral Arterial Disease
Keywords: Platelets; optical aggregometry; Lower Limb disease
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease | interventions — Clopidogrel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples With DNA — Blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Isolated coronary involvement (Group 1): Patients with previous infarction and isolated coronary involvement
  Interventions: Drug: Clopidogrel
- Concomitant presence of Lower Extremity Peripheral Artery Disease (Group 2): Patients with previous AMI and concomitant presence of Lower Extremity Peripheral Artery Disease
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 75 mg once a day for 14 days.

SUMMARY:
After an episode of acute ischemic syndrome, patients with concomitant peripheral arterial disease have a worse short- and long-term prognosis compared to patients with isolated coronary disease, but the mechanisms responsible are poorly understood. In this population, the presence of high platelet aggregability despite the use of antiplatelet drugs is related to a greater risk of future complications, including heart attack and death from all causes.

Thus, the main objective of the present project is to evaluate the role of platelet aggregability, analyzed by optical aggregometry using the AggRAM® equipment, in patients with a history of previous acute myocardial infarction with and without the presence of peripheral arterial disease. Among the secondary objectives, it is worth analyzing platelet aggregability, in both groups, using the Plateletworks® method. This is a case-control study, with groups differentiated by the presence or absence of peripheral arterial disease, matched by sex and age.

It is expected that, in the end, relevant aspects related to platelet aggregation will be better characterized in this high cardiovascular risk population, with a likely impact on new therapeutic strategies that can positively influence the morbidity and mortality of these patients.

DETAILED DESCRIPTION:
Polyvascular involvement is frequently present in atherosclerotic disease (AD). Lower Extremity Peripheral Artery Disease (PAD) represents one of the manifestations of AD; it is estimated that around 47% of people with atherosclerotic disease have involvement in more than one vascular bed, with coronary atherosclerotic disease and lower limb AD being the most prevalent.

Initial studies suggest that platelet aggregability is increased in patients with PAD and the level of platelet aggregability is associated with the severity of PAD.However, to our knowledge, there are no studies in the literature analyzing platelet aggregability in patients with previous AMI with and without the concomitant presence of PAD, which is the proposal of this research project.

This study is an observational, case-control study, matched by sex and age. Two groups will be selected: Patients with previous infarction and isolated coronary involvement (Group 1); Patients with previous AMI and concomitant presence of PAD of the lower limbs (Group 2).

Primary objective is compare platelet aggregability analyzed by optical aggregometry-ADP (AggRAM™- Helena Laboratories) between the groups. Secondary objetives includes laboratorial test of inflammation, coagulation and subgroup analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥ 18 years;
2. Daily use of AAS 81-100 mg and statins;
3. History of acute myocardial infarction, proven by medical record analysis;
4. Group 2 (patients with PAD): Ankle-Brachial Index number (ABI) ≤ 0.9 in at least one of the lower limbs. In diabetic patients with ABI > 1.4, the Hallux-Brachialis Index should be performed if possible; if the patient presents a value < 0.7, they can be included;
5. Signing of the Free and Informed Consent Form.

Exclusion Criteria:

1. Use of adenosine-diphosphate (ADP) receptor antagonists in the last 7 days before inclusion in the study;
2. Use of Anticoagulants in the last 30 days before inclusion in the study;
3. Clopidogrel allergy;
4. Known atherosclerotic carotid disease or carotid bruit;
5. History of upper gastrointestinal bleeding in the last 12 months;
6. Pregnancy or lactation;
7. Known platelet dysfunction or platelet count <100,000/µL or >450,000/µL;
8. Known liver disease or coagulation disorder;
9. Hematocrit less than 34% or greater than 55%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: Patients with previous infarction and isolated coronary involvement
  Group 2: Patients with previous AMI and concomitant presence of Lower Extremity Peripheral Artery Disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-05-13 (Estimated); Study Completion 2028-05-13 (Estimated)

PRIMARY OUTCOMES:
Aggregability analyzed by optical aggregometry-ADP (AggRAM™- Helena Laboratories) | 14 days
  Compare platelet aggregability analyzed by optical aggregometry-ADP (AggRAM™- Helena Laboratórios) between both groups

SECONDARY OUTCOMES:
Platelet aggregability by AggRAM™ arachidonic acid at baseline; | Baseline
  Avaliation of Platelet aggregability by AggRAM™ arachidonic acid at baseline;
Platelet aggregability by AggRAM™ ADP after 14 days of use of Clopidogrel 75 mg/day; | 14 days
  Evaluation of Platelet aggregability by AggRAM™ ADP after 14 days of use of Clopidogrel 75 mg/day;
Platelet aggregability by Plateletworks-ADP at baseline and after 14 days of use of Clopidogrel 75 mg/day; | 14 days
  Evaluation of Platelet aggregability by Plateletworks-ADP at baseline and after 14 days of use of Clopidogrel 75 mg/day;
Serum levels of ultrasensitive C-reactive protein (hs-CRP); | Baseline
  Avaliation of Serum levels of ultrasensitive C-reactive protein (hs-CRP)
Serum levels of immature platelets; | Baseline
  Evaluation of Serum levels of immature platelets;
Platelet count; | Baseline
  Evaluation of Platelet count;
Mean platelet volume (MPV); | Baseline
  Evaluation of Mean platelet volume (MPV);
Serum levels of P-Selectin ; | Baseline
  Evaluation of Serum levels of P-Selectin ;
Serum levels of type I plasminogen activator inhibitor (PAI 1); | Baseline
  Evaluation of Serum levels of type I plasminogen activator inhibitor (PAI 1);
Serum levels of interleukin 6; | Baseline
  Evaluation of Serum levels of interleukin 6;
Serum levels of Interleukin 1 | Baseline
  Evaluation of Serum levels of Interleukin 1
Serum levels of cholesterol ester transfer proteins; | Baseline
  Evaluation of Serum levels of cholesterol ester transfer proteins;
Serum levels of Lipoprotein(a) (LPa) | Baseline
  Evaluation of Serum levels of Lipoprotein(a) (LPa)

OTHER OUTCOMES:
Subgroup Analysis- Sex | Baseline and 14 days
  Sex (male/female)
Subgroup Analysis- Age | Baseline and 14 days
  Age (≥65 years or < 65 years)
Subgroup Analysis- hypertension | Baseline and 14 days
  History of arterial hypertension (presence or not);
Subgroup Analysis- BDI | Baseline and 14 days
  Body Mass Index (<30 or ≥ 30 kg/m2);
Subgroup Analysis- Diabetes mellitus | Baseline and 14 days
  Diabetes mellitus (presence or not);
Subgroup Analysis-Glomerular filtration rate | Baseline and 14 days
  Glomerular filtration rate (CKD EPI) (< 60ml/min/m2 or ≥ 60 ml/min/m2);
Subgroup Analysis- Smoking | Baseline and 14 days
  Current smoking (yes or no);
Subgroup Analysis- Ankle-brachial index number | Baseline and 14 days
  ABI 0.41-0.90 (mild/moderate) or <0.41 (Severe) or history of amputation.
Subgroup Analysis- Glycated hemoglobin | Baseline and 14 days
  Glycated hemoglobin(more or less than 8%);
Subgroup Analysis- Use of proton pump inhibitor | Baseline and 14 days
  Use of proton pump inhibitor (yes or no).

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute (InCor) / University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez Mejias EL, Faxas SM, Taveras NT, Talpur AS, Kumar J, Khalid M, Aruwani SK, Khalid D, Khalid H, Memon S. Peripheral Artery Disease as a Risk Factor for Myocardial Infarction. Cureus. 2021 Jun 15;13(6):e15655. doi: 10.7759/cureus.15655. eCollection 2021 Jun. PMID 34277248
- [Background] Hirsch AT, Criqui MH, Treat-Jacobson D, Regensteiner JG, Creager MA, Olin JW, Krook SH, Hunninghake DB, Comerota AJ, Walsh ME, McDermott MM, Hiatt WR. Peripheral arterial disease detection, awareness, and treatment in primary care. JAMA. 2001 Sep 19;286(11):1317-24. doi: 10.1001/jama.286.11.1317. PMID 11560536
- [Background] Bauersachs R, Zeymer U, Briere JB, Marre C, Bowrin K, Huelsebeck M. Burden of Coronary Artery Disease and Peripheral Artery Disease: A Literature Review. Cardiovasc Ther. 2019 Nov 26;2019:8295054. doi: 10.1155/2019/8295054. eCollection 2019. PMID 32099582
- [Background] Fox KA, Carruthers KF, Dunbar DR, Graham C, Manning JR, De Raedt H, Buysschaert I, Lambrechts D, Van de Werf F. Underestimated and under-recognized: the late consequences of acute coronary syndrome (GRACE UK-Belgian Study). Eur Heart J. 2010 Nov;31(22):2755-64. doi: 10.1093/eurheartj/ehq326. Epub 2010 Aug 30. PMID 20805110
- [Background] Nicolau JC, Bhatt DL, Roe MT, Lokhnygina Y, Neely B, Corbalan R, Leiva-Pons JL, Martinez F, Goodman SG, Winters KJ, Verheugt FW, Armstrong PW, White HD, Fox KA, Prabhakaran D, Ohman EM; TRILOGY ACS investigators. Concomitant proton-pump inhibitor use, platelet activity, and clinical outcomes in patients with acute coronary syndromes treated with prasugrel versus clopidogrel and managed without revascularization: insights from the Targeted Platelet Inhibition to Clarify the Optimal Strategy to Medically Manage Acute Coronary Syndromes trial. Am Heart J. 2015 Oct;170(4):683-694.e3. doi: 10.1016/j.ahj.2015.05.017. Epub 2015 Jun 11. PMID 26386792
- [Background] Nicolau JC, Feitosa Filho GS, Petriz JL, Furtado RHM, Precoma DB, Lemke W, Lopes RD, Timerman A, Marin Neto JA, Bezerra Neto L, Gomes BFO, Santos ECL, Piegas LS, Soeiro AM, Negri AJA, Franci A, Markman Filho B, Baccaro BM, Montenegro CEL, Rochitte CE, Barbosa CJDG, Virgens CMBD, Stefanini E, Manenti ERF, Lima FG, Monteiro Junior FDC, Correa Filho H, Pena HPM, Pinto IMF, Falcao JLAA, Sena JP, Peixoto JM, Souza JA, Silva LSD, Maia LN, Ohe LN, Baracioli LM, Dallan LAO, Dallan LAP, Mattos LAPE, Bodanese LC, Ritt LEF, Canesin MF, Rivas MBDS, Franken M, Magalhaes MJG, Oliveira Junior MT, Filgueiras Filho NM, Dutra OP, Coelho OR, Leaes PE, Rossi PRF, Soares PR, Lemos Neto PA, Farsky PS, Cavalcanti RRC, Alves RJ, Kalil RAK, Esporcatte R, Marino RL, Giraldez RRCV, Meneghelo RS, Lima RSL, Ramos RF, Falcao SNDRS, Dalcoquio TF, Lemke VMG, Chalela WA, Mathias Junior W. Brazilian Society of Cardiology Guidelines on Unstable Angina and Acute Myocardial Infarction without ST-Segment Elevation - 2021. Arq Bras Cardiol. 2021 Jul;117(1):181-264. doi: 10.36660/abc.20210180. No abstract available. English, Portuguese. PMID 34320090
- [Background] Smolina K, Wright FL, Rayner M, Goldacre MJ. Long-term survival and recurrence after acute myocardial infarction in England, 2004 to 2010. Circ Cardiovasc Qual Outcomes. 2012 Jul 1;5(4):532-40. doi: 10.1161/CIRCOUTCOMES.111.964700. Epub 2012 Jun 26. PMID 22740013
- [Background] Steen DL, Khan I, Andrade K, Koumas A, Giugliano RP. Event Rates and Risk Factors for Recurrent Cardiovascular Events and Mortality in a Contemporary Post Acute Coronary Syndrome Population Representing 239 234 Patients During 2005 to 2018 in the United States. J Am Heart Assoc. 2022 May 3;11(9):e022198. doi: 10.1161/JAHA.121.022198. Epub 2022 Apr 27. PMID 35475346
- [Background] Nakatani D, Sakata Y, Suna S, Usami M, Matsumoto S, Shimizu M, Sumitsuji S, Kawano S, Ueda Y, Hamasaki T, Sato H, Nanto S, Hori M, Komuro I; Osaka Acute Coronary Insufficiency Study (OACIS) Investigators. Incidence, predictors, and subsequent mortality risk of recurrent myocardial infarction in patients following discharge for acute myocardial infarction. Circ J. 2013;77(2):439-46. doi: 10.1253/circj.cj-11-1059. Epub 2012 Oct 17. PMID 23075765
- [Background] Thune JJ, Signorovitch JE, Kober L, McMurray JJ, Swedberg K, Rouleau J, Maggioni A, Velazquez E, Califf R, Pfeffer MA, Solomon SD. Predictors and prognostic impact of recurrent myocardial infarction in patients with left ventricular dysfunction, heart failure, or both following a first myocardial infarction. Eur J Heart Fail. 2011 Feb;13(2):148-53. doi: 10.1093/eurjhf/hfq194. Epub 2010 Oct 29. PMID 21037250
- [Background] Attar R, Wester A, Koul S, Eggert S, Andell P. Peripheral artery disease and outcomes in patients with acute myocardial infarction. Open Heart. 2019 May 12;6(1):e001004. doi: 10.1136/openhrt-2018-001004. eCollection 2019. PMID 31245013
- [Background] Patel MR, Becker RC, Wojdyla DM, Emanuelsson H, Hiatt WR, Horrow J, Husted S, Mahaffey KW, Steg PG, Storey RF, Wallentin L, James SK. Cardiovascular events in acute coronary syndrome patients with peripheral arterial disease treated with ticagrelor compared with clopidogrel: Data from the PLATO Trial. Eur J Prev Cardiol. 2015 Jun;22(6):734-42. doi: 10.1177/2047487314533215. Epub 2014 May 15. PMID 24830710
- [Background] Akahori H, Masuyama T, Imanaka T, Nakao K, Ozaki Y, Kimura K, Ako J, Noguchi T, Suwa S, Fujimoto K, Nakama Y, Morita T, Shimizu W, Saito Y, Hirohata A, Morita Y, Inoue T, Okamura A, Mano T, Hirata K, Tanabe K, Shibata Y, Owa M, Tsujita K, Funayama H, Kokubu N, Kozuma K, Uemura S, Tobaru T, Saku K, Oshima S, Nishimura K, Miyamoto Y, Ogawa H, Ishihara M; J-MINUET investigators. Impact of peripheral artery disease on prognosis after myocardial infarction: The J-MINUET study. J Cardiol. 2020 Oct;76(4):402-406. doi: 10.1016/j.jjcc.2020.05.014. Epub 2020 Jun 9. PMID 32532585
- [Background] Andersen P, Kragholm K, Torp-Pedersen C, Jensen SE, Attar R. The impact of peripheral artery disease on major adverse cardiovascular events following myocardial infarction. Int J Cardiol. 2021 Nov 15;343:131-137. doi: 10.1016/j.ijcard.2021.08.053. Epub 2021 Sep 6. PMID 34499974
- [Background] Breet NJ, van Werkum JW, Bouman HJ, Kelder JC, Ruven HJ, Bal ET, Deneer VH, Harmsze AM, van der Heyden JA, Rensing BJ, Suttorp MJ, Hackeng CM, ten Berg JM. Comparison of platelet function tests in predicting clinical outcome in patients undergoing coronary stent implantation. JAMA. 2010 Feb 24;303(8):754-62. doi: 10.1001/jama.2010.181. PMID 20179285
- [Background] Cassar K, Bachoo P, Ford I, Greaves M, Brittenden J. Platelet activation is increased in peripheral arterial disease. J Vasc Surg. 2003 Jul;38(1):99-103. doi: 10.1016/s0741-5214(03)00129-0. PMID 12844097
- [Background] Robless PA, Okonko D, Lintott P, Mansfield AO, Mikhailidis DP, Stansby GP. Increased platelet aggregation and activation in peripheral arterial disease. Eur J Vasc Endovasc Surg. 2003 Jan;25(1):16-22. doi: 10.1053/ejvs.2002.1794. PMID 12525806
- [Background] Galt SW, McDaniel MD, Ault KA, Mitchell J, Cronenwett JL. Flow cytometric assessment of platelet function in patients with peripheral arterial occlusive disease. J Vasc Surg. 1991 Dec;14(6):747-55; discussion 755-6. doi: 10.1067/mva.1991.33419. PMID 1720468
- [Background] Rajagopalan S, Mckay I, Ford I, Bachoo P, Greaves M, Brittenden J. Platelet activation increases with the severity of peripheral arterial disease: implications for clinical management. J Vasc Surg. 2007 Sep;46(3):485-90. doi: 10.1016/j.jvs.2007.05.039. PMID 17826235